CLINICAL TRIAL: NCT02323126
Title: A Phase II, Multicenter, Open-label Study of EGF816 in Combination With Nivolumab in Adult Patients With EGFR Mutated Non-small Cell Lung Cancer and of INC280 in Combination With Nivolumab in Adult Patients With cMet Positive Non-small Cell Lung Cancer
Brief Title: Study of Efficacy and Safety of Nivolumab in Combination With EGF816 and of Nivolumab in Combination With INC280 in Patients With Previously Treated Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to low patient recruitment caused by the change in the treatment landscape of NSCLC.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEGF816X2201C; 2014-003731-20 (EudraCT Number)
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; NSCLC; EGFR-mutated; EGF816; INC280; Nivolumab; EGFR-T790M NSCLC; EGFR wild-type (wt); cMET positive NSCLC; cMET negative NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nazartinib; capmatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab and EGF816 (Experimental): Group 1: EGF816 150 mg QD + Nivolumab 3 mg/kg Q2W
  Interventions: Drug: EGF816; Drug: Nivolumab
- Nivolumab and INC280, high cMet (Experimental): Group 2A: INC280 400 mg BID, High cMET + Nivolumab 3 mg/kg Q2W
  Interventions: Drug: INC280; Drug: Nivolumab
- Nivolumab and INC280, low cMet (Experimental): Group 2B: INC280 400 mg BID, Low cMet + Nivolumab 3 mg/kg Q2W
  Interventions: Drug: INC280; Drug: Nivolumab

INTERVENTIONS:
Drug: EGF816 — EGF816 150 mg once daily (QD) administered orally as a capsule
  Arms: Nivolumab and EGF816
Drug: INC280 — INC280 400 mg twice daily (BID) administered orally as a tablet
  Arms: Nivolumab and INC280, high cMet; Nivolumab and INC280, low cMet
Drug: Nivolumab — Nivolumab 3 mg/kg every 2 weeks (Q2W) administered by intravenous infusion

SUMMARY:
To determine the efficacy and safety of nivolumab in combination with EGF816 and of nivolumab in combination with INC280 in previously treated NSCLC patients

DETAILED DESCRIPTION:
This was a phase II, multi-center, open-label study in patients with advanced non-small cell lung cancer (NSCLC). Patients were allocated based on their epidermal growth factor receptor (EGFR) status to one of the 2 groups: Group 1 - EGFR T790M NSCLC treated with EGF816 150 mg once daily (QD) + nivolumab 3 mg/kg every 2 weeks (Q2W), and Group 2 - EGFR wild type (wt) NSCLC treated with INC280 400 mg twice daily (BID) + nivolumab 3 mg/kg Q2W. Patients in Group 2 were subdivided into 2 subgroups based on c-Mesenchymal-epithelial transition (cMet) status: Subgroup A - high cMet (referred to as Group 2A) and Subgroup B- low cMet (referred to as Group 2B).

Patients could continue study treatment until patients experienced unacceptable toxicity that precluded any further treatment, disease progression and/or treatment was discontinued at the discretion of the investigator or withdrawal of consent, or the patient was transferred to a Novartis roll-over study or an alternative treatment option that could continue to provide study treatments. Following the approval of a protocol amendment, the maximum treatment duration for nivolumab could not exceed 2 years and patients who had received nivolumab beyond 2 years were discontinued from nivolumab treatment and continued on EGF816 or INC280 alone.

The primary objective of the trial was to estimate the clinical activity of nivolumab in combination with EGF816 or INC280.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures
* Presence of at least one measurable lesion according to RECIST v.1.1
* ECOG performance status ≤ 2
* Patients with histologically documented locally advanced, recurrent and/or metastatic NSCLC
* Tumor tissue for determination and/or confirmation of genetic pre-requisites (i.e. EGFR T790M positivity post progression on EGFR TKI for Group 1; cMet status for Group 2) must be provided for analysis

Group 1 patients:

* Patients with EGFR T790M NSCLC (adenocarcinoma)
* Documented progression of disease according to RECIST v1.1 following primary standard of care (e.g. erlotinib, gefitinib)

Group 2 patients:

* Patients with EGFR wild-type NSCLC
* Documented progression of disease according to RECIST v1.1 following standard of care (e.g. platinum doublet).

Exclusion Criteria:

* Patients who have received more than one prior line of EGFR TKI therapy1 (applies only to Group 1)
* Previous treatment with a c-MET inhibitor or HGF-targeting therapy (applies only to Group 2)
* Patients with brain metastases. However, if radiation therapy and/or surgery has been completed and serial evaluation by CT (with contrast enhancement) or MRI over a minimum of one month demonstrates the disease to be stable and if the patient remains asymptomatic without the need for treatment with steroids
* Patients who require emergent use of systemic steroids, chronic use of prednisone (greater than 10mg or an equivalent steroid dose daily) or emergent surgery and/or radiotherapy.
* History of allergy or hypersensitivity to nivolumab components
* Patients with any known or suspected, current or past history of, autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients with a condition requiring chronic systemic treatment with either corticosteroids(> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of treatment start. Inhaled or topical steroids, and adrenal replacement steroid doses> 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Patients who have been treated with prior PD-1 and PD-L1 agents
* Patients who previously received agents targeting c-MET and/or EGFR T790M Note: Previous treatment with afatinib may be allowable after discussions between Novartis and Investigator.
* Patients with the following laboratory abnormalities:

  * Absolute Neutrophil Count (ANC) <1.5 x 109/L
  * Hemoglobin (Hgb) <9 g/dL
  * Platelets <100 x 109/L
  * Total bilirubin >1.5 x upper limit of normal (ULN). For patients with Gilbert's syndrome total bilirubin >2.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3 x ULN
  * Serum creatinine >1.5 x ULN and/or measured or calculated creatinine clearance <75% LLN
  * For patients being screened for Group 2, asymptomatic serum amylase > CTCAE Grade 2 (1.5-2.0 x ULN). Patients with Grade 1 or Grade 2 serum amylase at the beginning of the study must be confirmed to have no signs or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
  * For patients being screened for Group 2: Serum lipase > ULN
* Female patients who are either pregnant or nursing.
* Women of child bearing potential who refuse or are not able to use a highly effective method of contraception as defined in the study protocol.
* Sexually active males unless they use a condom during intercourse while taking drug and for 31 weeks after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- University of Texas MD Anderson Cancer Center Thoractic Head/Neck Med.Onc(2), Houston, Texas, United States
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Chermside, Queensland
- Novartis Investigative Site, La Tronche, France
- Novartis Investigative Site, Cologne, North Rhine-Westphalia, Germany
- Italy (2):
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Aviano, PN
- Novartis Investigative Site, Singapore, Singapore
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Chur, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Felip E, Metro G, Tan DSW, Wolf J, Mark M, Boyer M, Hughes BGM, Bearz A, Moro-Sibilot D, Le X, Puente J, Massuti B, Tiedt R, Wang Y, Xu C, Mardjuadi FI, Cobo M. Capmatinib plus nivolumab in pretreated patients with EGFR wild-type advanced non-small cell lung cancer. Lung Cancer. 2024 Jun;192:107820. doi: 10.1016/j.lungcan.2024.107820. Epub 2024 May 10. PMID 38763104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 13 investigative sites in 8 countries.
Pre-assignment Details: All patients were required to sign the molecular pre-screening consent to allow for the collection and submission of tumor tissue for determination and/or confirmation of protocol specific pre-requisite genetic alterations. After the molecular pre-screening, the screening period began once patients had signed the study informed consent. Screening evaluations were performed within 28 days prior to the first dose of study medication. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Started | 18 | 16 | 30
Completed | 0 | 0 | 0
Not Completed | 18 | 16 | 30
Not completed — Patient / guardian decision | 0 | 1 | 2
Not completed — Progressive disease | 14 | 8 | 14
Not completed — Physician Decision | 0 | 1 | 3
Not completed — Death | 1 | 1 | 4
Not completed — Adverse Event | 3 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet | Total
Number analyzed (Participants) | 18 | 16 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.77) | 63.8 (13.05) | 64.9 (8.45) | 64.0 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 15 | 35
  Male | 6 | 8 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 2 | 7
  Caucasian | 14 | 14 | 26 | 54
  Other | 0 | 0 | 1 | 1
  Unknown | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate at 6 Months Per RECIST v1.1
Description: PFS rate represents the percentage of participants without a first documented progression or death due to any cause after the start of study treatment. Tumor response was based on local investigator assessment as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
  PFS was modeled using a Weibull distribution and the PFS rate at 6 months was estimated from the posterior distribution.
Time Frame: 6 months
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
percentage of participants | 63.4 [45.7 to 79.2] | 68.9 [48.5 to 85.7] | 50.9 [35.6 to 66.4]

2. Secondary Outcome: Overall Response Rate (ORR) Per RECIST v1.1
Description: Tumor response was based on local investigator assessment as per RECIST v1.1. ORR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until end of treatment, assessed up to 4.7 years
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
Participants | 7 | 4 | 5

3. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1
Description: Tumor response was based on local investigator assessment as per RECIST v1.1. DCR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Time Frame: From start of treatment until end of treatment, assessed up to 4.7 years
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
Participants | 17 | 13 | 13

4. Secondary Outcome: Median Progression-Free Survival (PFS) Per RECIST v1.1
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment. The median PFS was estimated using the Kaplan-Meier method.
  Tumor response was based on local investigator assessment as per RECIST v1.1
Time Frame: From start of treatment to first documented progression or death, assessed up to 5 years
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
months | 7.4 [3.7 to 11.1] | 6.2 [3.5 to 19.2] | 4.2 [1.8 to 7.4]

5. Secondary Outcome: Progression-Free Survival (PFS) Rate at 3 Months Per RECIST v1.1
Description: PFS rate represents the percentage of participants without a first documented progression or death due to any cause after the start of study treatment. Tumor response was based on local investigator assessment as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
  The PFS rate at 3 months was estimated using the Kaplan-Meier method.
Time Frame: 3 months
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
percentage of participants | 83.3 [56.8 to 94.3] | 86.7 [56.4 to 96.5] | 53.8 [33.3 to 70.6]

6. Secondary Outcome: Overall Survival (OS) at 1 Year
Description: OS represents the percentage of participants who are alive after the start of study treatment. OS at 1 year was estimated using the Kaplan-Meier method.
Time Frame: 1 year
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
percentage of participants | 55.6 [30.5 to 74.8] | 72.3 [41.5 to 88.7] | 32.5 [15.8 to 50.5]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose of study medication up to 100 days after last dose of study medication, with a maximum duration of 5 years
Population: All patients who had received at least 1 dose of INC280, EGF816 or nivolumab and had at least 1 valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
Participants
  AEs | 18 | 16 | 30
  Treatment-related AEs | 17 | 16 | 27
  AEs with grade 3/4 | 18 | 14 | 24
  Treatment-related AEs with grade 3/4 | 13 | 12 | 16
  SAEs | 14 | 8 | 18
  Treatment-related SAEs | 6 | 4 | 7
  Fatal SAEs | 4 | 1 | 4
  Treatment related fatal SAEs | 2 | 0 | 0
  AEs leading to discontinuation | 5 | 7 | 11
  Treatment-related AEs leading to discontinuation | 5 | 7 | 9
  AEs leading to dose adjustment/interruption | 15 | 14 | 23

8. Secondary Outcome: Number of Participants With Dose Reductions and Dose Interruptions of EGF816, INC280 and Nivolumab
Description: Number of participants with at least one dose reduction of EGF816, INC280 or nivolumab and number of participants with at least one dose interruption of EGF816, INC280 or nivolumab.
  Dose reduction was not allowed for nivolumab in this study.
Time Frame: From first dose of study treatment until last dose of study treatment, up to maximum 4.7 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
Participants
  EGF816, dose reduction: number analyzed (Participants) | 18 | 0 | 0
  EGF816, dose reduction | 5 |  |
  EGF816, dose interruption: number analyzed (Participants) | 18 | 0 | 0
  EGF816, dose interruption | 14 |  |
  INC280, dose reduction: number analyzed (Participants) | 0 | 16 | 30
  INC280, dose reduction |  | 7 | 10
  INC280, dose interruption: number analyzed (Participants) | 0 | 16 | 30
  INC280, dose interruption |  | 14 | 25
  Nivolumab, dose reduction | 0 | 0 | 0
  Nivolumab, dose interruption | 12 | 10 | 15

9. Secondary Outcome: Dose Intensity of EGF816 and INC280
Description: Dose intensity (mg/day) of EGF816 and INC280 was calculated as actual cumulative dose in milligrams divided by duration of exposure in days.
Time Frame: From first dose of study treatment until last dose of study treatment, up to maximum 4.7 years
Population: as for outcome 7
Measure: Median (Full Range); unit: mg/day
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
mg/day
  EGF816: number analyzed (Participants) | 18 | 0 | 0
  EGF816 | 141.5 [81 to 150] |  |
  INC280: number analyzed (Participants) | 0 | 16 | 30
  INC280 |  | 609.4 [254 to 800] | 636.7 [240 to 800]

10. Secondary Outcome: Dose Intensity of Nivolumab
Description: Dose intensity (mg/kg biweekly) of nivolumab was calculated as actual cumulative dose in mg/kg divided by duration of exposure in days and then multiplied by 14 days (2 weeks).
Time Frame: From first dose of study treatment until last dose of study treatment, up to maximum 4.7 years
Population: as for outcome 7
Measure: Median (Full Range); unit: mg/kg/2-week
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 16 | 30
mg/kg/2-week | 3.0 [3 to 3] | 3.0 [3 to 3] | 3.0 [3 to 3]

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post EGF816 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: All patients who had extensive PK sampling and provided an EGF816 evaluable PK profile on Cycle 1 Day 15. The EGF816 PK profile was considered evaluable if all the following conditions were satisfied: patient had received planned doses and patient had provided at least 1 valid primary PK parameter (Cmax, Tmax, AUClast).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nivolumab and EGF816
Number analyzed (Participants) | 11
ng/mL | 935 (40.8)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post EGF816 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Nivolumab and EGF816
Number analyzed (Participants) | 11
hours | 3.00 [1.00 to 6.00]

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post EGF816 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Nivolumab and EGF816
Number analyzed (Participants) | 11
hr*ng/mL | 5560 (42.8)

14. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods. Cmin is defined as the minimum observed plasma concentration following a dose.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post EGF816 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nivolumab and EGF816
Number analyzed (Participants) | 11
ng/mL | 398 (48.8)

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post INC280 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: All patients who had extensive PK sampling and provided an INC280 evaluable PK profile on Cycle 1 Day 15. The INC280 PK profile was considered evaluable if all the following conditions were satisfied: patient had received planned doses and patient had provided at least 1 valid primary PK parameter (Cmax, Tmax, AUClast). In the Group 2B, no patients provided an INC280 evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 5 | 0
ng/mL | 6190 (83.9) |

16. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post INC280 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 5 | 0
hours | 0.983 [0.667 to 1.08] |

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post INC280 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 5 | 0
hr*ng/mL | 19300 (97.5) |

18. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Cmin is defined as the minimum observed plasma concentration following a dose.
Time Frame: pre-dose, 1, 3, 6 and 8 hours post INC280 dose on Cycle 1 Day 15. The duration of one cycle was 28 days.
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 5 | 0
ng/mL | 428 (105) |

19. Secondary Outcome: Pre-dose Serum Concentration of Nivolumab
Description: Nivolumab serum concentrations were assessed in samples taken at pre-dose. Pre-dose samples were collected before the next dose administration.
Time Frame: pre-dose on Cycle 1 Day 1 (groups 2A and 2B only) and pre-dose on Cycle 1 Day 15 and Cycle 2 Day 1 (all groups). The duration of one cycle was 28 days.
Population: All patients who had provided at least 1 evaluable nivolumab PK concentration. For a nivolumab PK concentration to be evaluable in pre-dose samples, a patient was required to have the sample collected before the next dose administration. Samples were not collected in Group 1 on Cycle 1 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet
Number analyzed (Participants) | 18 | 15 | 29
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 7 | 16
  Cycle 1 Day 1 |  | NA (NA) — Concentrations below the limit of quantification (<0.20 ng/mL) | NA (NA) — Concentrations below the limit of quantification (<0.20 ng/mL)
  Cycle 1 Day 15: number analyzed (Participants) | 17 | 13 | 23
  Cycle 1 Day 15 | 17.2 (28.6) | 18.6 (45.3) | 19.5 (35.6)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 10 | 22
  Cycle 2 Day 1 | 21.3 (54.6) | 35.7 (26.6) | 26.4 (77.1)

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to 100 days after last dose of study medication, with a maximum duration of 5 years.
Description: Any sign or symptom that occurs during the study treatment plus 100 days after last dose.
Groups:
- Nivolumab and INC280, High+Low cMet: Group 2A+2B (low and high cMet): INC280 400 mg BID + Nivolumab 3 mg/kg Q2W
Arm/Group | Nivolumab and EGF816 | Nivolumab and INC280, High cMet | Nivolumab and INC280, Low cMet | Nivolumab and INC280, High+Low cMet
All-Cause Mortality (participants affected / at risk) | 8/18 | 4/16 | 10/30 | 14/46
Serious Adverse Events (participants affected / at risk) | 14/18 | 8/16 | 18/30 | 26/46
Other Adverse Events (participants affected / at risk) | 18/18 | 16/16 | 29/30 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and EGF816 (N=18) | Nivolumab and INC280, High cMet (N=16) | Nivolumab and INC280, Low cMet (N=30) | Nivolumab and INC280, High+Low cMet (N=46)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Condition aggravated (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 3 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Giant cell arteritis (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and EGF816 (N=18) | Nivolumab and INC280, High cMet (N=16) | Nivolumab and INC280, Low cMet (N=30) | Nivolumab and INC280, High+Low cMet (N=46)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 7 | 11
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 2
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 0 | 2
Hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 2
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3 | 4
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 6 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 5 | 13 | 12 | 25
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 2 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9 | 7 | 16
Asthenia (General disorders) | 7 | 6 | 10 | 16
Catheter site swelling (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 5 | 4 | 9
Gait disturbance (General disorders) | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 2
Oedema (General disorders) | 0 | 1 | 1 | 2
Oedema peripheral (General disorders) | 1 | 8 | 8 | 16
Pain (General disorders) | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 1 | 2 | 0 | 2
Pyrexia (General disorders) | 10 | 6 | 3 | 9
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 1
Pulpitis dental (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 5 | 7
Amylase increased (Investigations) | 6 | 9 | 6 | 15
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 5 | 6
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 6 | 6
Blood creatinine increased (Investigations) | 0 | 6 | 9 | 15
Blood glucose increased (Investigations) | 0 | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 0 | 3
Lipase increased (Investigations) | 4 | 7 | 6 | 13
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2 | 2
Transaminases increased (Investigations) | 0 | 1 | 2 | 3
Weight decreased (Investigations) | 3 | 2 | 2 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 2
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 9 | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 9 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 7 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Infected naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 4
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 5 | 0 | 5
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 2
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Device occlusion (Product Issues) | 0 | 1 | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 2 | 1 | 3
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Perineal fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 7 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 12 | 3 | 4 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Giant cell arteritis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT02323126/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02323126/SAP_002.pdf